CLINICAL TRIAL: NCT00203424
Title: A Phase II Trial of Adjuvant Bevacizumab and Erlotinib in Patients at High Risk for Early Relapse Following Radical Prostatectomy for Prostate Cancer
Brief Title: Treatment of Prostate Cancer With Adjuvant Bevacizumab Plus Erlotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORI GU-01; 05-07-102 (Other: UCLA IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + Bevacizumab (Experimental): Participants received Erlotinib every day for 24 weeks and Bevacizumab every 3 weeks for a total of 8 doses
  Interventions: Drug: Erlotinib + Bevacizumab

INTERVENTIONS:
Drug: Erlotinib + Bevacizumab — Erlotinib every day for 24 weeks and Bevacizumab every 3 weeks for a total of 8 doses

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of bevacizumab plus erlotinib following radical prostatectomy.

DETAILED DESCRIPTION:
This study explores the anti-tumor activity of adjuvant bevacizumab plus erlotinib in a select group of prostate cancer patients deemed at high risk for early relapse following radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of > 80
* Patients must have localized, organ-confined prostate cancer documented by physical examination, CT scan, or bone scan, and must have undergone radical prostatectomy. Post RP must have documented node negative prostate cancer.
* Pretreatment granulocyte count > 1500/mm3, hemoglobin > 9.0 g/dL, and platelet count > 100,000/mm3,
* Normal PT and PTT
* Serum creatinine < 2.0 mg/dL
* Adequate hepatic function with a serum bilirubin < upper limit of normal (ULN), AST and ALT < 1.5x ULN, and alkaline phosphatase < 2.5x ULN.
* High-risk prostate cancer defined as a pre-RP prostate specific antigen level > 15 ng/dL or a Gleason score of > 8 or Stage T3 disease or positive surgical margins
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for 3 months thereafter

Exclusion Criteria:

* Evidence of small cell (neuroendocrine) tumor
* Evidence of metastatic disease
* Prior administration of immunotherapy, biological therapy, hormonal therapy or radiation therapy for prostate cancer
* Active secondary malignancies (other than basal cell carcinoma of the skin)
* Serious, nonhealing wound, ulcer, or bone fracture.
* Clinically significant cardiovascular disease (e.g., blood pressure of >150/100 mmHg, myocardial infarction, or unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or clinically significant peripheral vascular disease. Patients with a history of myocardial infarction or stroke within the last 6 months will be excluded.
* Presence of seizures not controlled with standard medical therapy
* Active infection requiring parenteral antibiotics at the time of the first administration of study drugs
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0.
* Current, recent (within the 4 weeks preceding Day 0), or planned participation in another experimental drug study
* Inability to comply with the study visit and follow-up schedule or procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Urine protein:creatinine ration > 1.0 at screening
* Evidence of bleeding diathesis or coagulopathy.
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 28 days prior to Day 0.
* Presence of central nervous system or brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz Kabbinavar, MD, Study Chair — Chief Medical Officer, TORI
Locations (16):
- United States (16):
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - San Diego Cancer Center, Vista, California
  - Cancer Institute of Florida, P.A., Orlando, Florida
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - South Texas Oncology and Hematology, P.A., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 6/23/2005 - 03/10/2009 Types of location: Academic medical clinics and community medical clinics.
Pre-assignment Details: There are no pre-assignment details to describe.
Groups:
- Erlotinib + Bevacizumab: 27 participants were screened for the study. 4 did not meet eligibility criteria,23 were registered to treatment period. 1 withdrew consent a day after registration and did not initiate study treatment.22 participants entered treatment period. Participants received Erlotinib every day for 24 weeks and Bevacizumab every 3 weeks for a total of 8 doses. The protocol instructed that pts be treated for 6 cycles. Of the 22 pts that started treatment, 11 completed the 6 cycles and the other 11 had to stop treatment prior to administration of 6th cycle. Of the 11 pts that did not complete all 6 cycles, 5 stopped treatment due to adverse event and were entered into the follow-up period. The 6 that stopped treatment due to withdrawal of consent and progressive disease did not enter the follow-up period. So 11 pts that completed 6 cycles of treatment plus 5 pts that did not complete 6 cycles of treatment due to an adverse event gives a total of 16 patients who entered follow-up period.
Period: Treatment Period
Arm/Group | Erlotinib + Bevacizumab
Started | 22 (23 subjects registered for treatment, 1 withdrew consent after registration,22 received treatment.)
Completed | 11 (Of 11 pts that did not complete treatment,5 stopped due to adverse event and entered followup period)
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 5
Not completed — progressive disease | 2
Period: Follow-up Period
Arm/Group | Erlotinib + Bevacizumab
Started | 16 (followup includes 11 pts that completed treatment + 5 pts who stopped treatment due to adverse event)
Completed | 10
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — progressive disease | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib + Bevacizumab: Participants that entered treatment period.
Arm/Group | Erlotinib + Bevacizumab
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 67 [51 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Bevacizumab Plus Erlotinib
Time Frame: Determined by time to tumor recurrence, as measured by rising prostate specific antigen (PSA) after radical prostatectomy.
Population: Of the 23 subjects registered for treatment, 19 were analysed for efficacy, 4 subjects were excluded from analysis because of withdrawal of subjects prior to first tumor assessment.
Measure: Number; unit: participants
Arm/Group | Bevacizumab+Erlotinib
Number analyzed (Participants) | 19
participants
  completed study without tumor progression | 9
  lost to follow-up unaffected by tumor recurrence | 1
  withdrawal by subjects unaffected by recurrence | 2
  affected by tumor recurrence | 7

2. Secondary Outcome: Time to Tumor Progression.
Description: Measured once for participants who experienced tumor recurrence per protocol. Imaging done to measure tumor progression only after documented tumor recurrence
Time Frame: Tumor progression assessed every 3 months during Follow-up Period for a maximum of 3 years after administration of first study treatment
Measure: Number; unit: days
Arm/Group | Bevacizumab+Erlotinib
Number analyzed (Participants) | 1
days | 314

3. Primary Outcome: Time to Tumor Recurrence
Time Frame: as for outcome 2
Measure: Mean (Full Range); unit: days
Arm/Group | Bevacizumab+Erlotinib
Number analyzed (Participants) | 7
days | 285 [42 to 835]

4. Secondary Outcome: Overall Survival
Time Frame: Survival status was assessed every 3 months after completion of study treatment for a maximum of 3 years after administration of first study treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab+Erlotinib
Number analyzed (Participants) | 22
participants
  Deceased | 0
  Alive | 15
  Lost to Follow-up | 1
  Withdrawal by subject | 6

ADVERSE EVENTS:
Time Frame: Adverse event (AE)data collected between 11/30/2005 and 1/26/2011. Therefore AE reporting period is 5.16 years or 5 years and 2 months, approximately.
Description: Systemic adverse event assessment occurred every 21 days through investigator assessment during Treatment Period and every 3 months during Follow-up Period.
Arm/Group | Erlotinib + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Bevacizumab (N=22)
Grade 3 hypertension related to bevacizumab (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Bevacizumab (N=22)
rash (Skin and subcutaneous tissue disorders) | 16
Fatigue (Musculoskeletal and connective tissue disorders) | 15
Diarrhea (Gastrointestinal disorders) | 14
Acne (Skin and subcutaneous tissue disorders) | 10
Hypertension (Cardiac disorders) | 9
Pain (General disorders) | 8
cough (Respiratory, thoracic and mediastinal disorders) | 8
Pruritis (Skin and subcutaneous tissue disorders) | 7
Epistaxis (Blood and lymphatic system disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 5
Infection (Infections and infestations) | 5
edema, limb (Blood and lymphatic system disorders) | 5
fever (General disorders) | 4
Anorexia (Gastrointestinal disorders) | 4
hemarrhoids (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 4
dry skin (Skin and subcutaneous tissue disorders) | 3
taste alteration (Gastrointestinal disorders) | 3
proteinuria (Metabolism and nutrition disorders) | 3
mood alteration (Nervous system disorders) | 3
headache (General disorders) | 3
chills (General disorders) | 2
cold symptoms (General disorders) | 2
insomnia (General disorders) | 2
peeling skin (Skin and subcutaneous tissue disorders) | 2
constipation (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 2
rectal bleeding (Vascular disorders) | 2
AST elevated (Metabolism and nutrition disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 2
serum total protein, decreased (Metabolism and nutrition disorders) | 2
neuropathy (Nervous system disorders) | 2
dysuria (General disorders) | 2
throat sore (General disorders) | 2
voice changes (Respiratory, thoracic and mediastinal disorders) | 2
urinary frequency, increased (Renal and urinary disorders) | 2
urinary retention (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
This was a small study with only 22 participants who received study treatment. With such a small sample size the study doesnt have the statistcical power to make categorical assessments or statements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The obligations of confidentiality shall apply for a period of 5 years beyond termination of Agreement between Sponsor and PI,but do not apply to the extent information:is or later becomes generally known to the public;is obtained from third party without restriction who had legal right to disclose;is already possessed by PI,as demonstrated by recipient's written records predating receipt from Sponsor;or is required to be disclosed pursuant to a subpoena,law,regulation,or other legal proceeding.